CLINICAL TRIAL: NCT00961246
Title: Web-Based Active Balance Childhood Study in Chinese-American (Web ABC Study): A Randomized Clinical Trial
Brief Title: Web-Based Active Balance Childhood Study in Chinese-American
Acronym: WEBABC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H11584-31742; KL2RR024130 (NIH)
Record Dates: First submitted 2009-08-16; First posted 2009-08-18 (Estimated); Last update posted 2013-09-25 (Estimated); Status verified 2013-09

CONDITIONS: Healthy
Keywords: web based intervention; individually-tailored; Chinese-American children; compared the changes in physical activity level; changes in dietary intake; changes in coping strategy used; changes in BMI

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- general health information group (Active Comparator): participants received general health information
  Interventions: Behavioral: general health information
- individually-tailored intervention (Experimental): participants received individually-tailored intervention
  Interventions: Behavioral: individually-tailored intervention

INTERVENTIONS:
Behavioral: general health information — participants received general health information
  Arms: general health information group
Behavioral: individually-tailored intervention — participants received individually-tailored intervention
  Arms: individually-tailored intervention

SUMMARY:
This study compares the feasibility and efficacy of an individually tailored, child-centered, Internet-based behavioral intervention with that of general Internet-based health information for improving health behaviors and relative weight in Chinese-American children during a 6-month period. A total of 60 children (age 10-14) and their families will be randomized to either the intervention group or control group. The intervention is based on the Social Cognitive Theory and Transtheoretical Model.

DETAILED DESCRIPTION:
The proposed study will use a randomized experimental design to examine the effects of an individually tailored, Internet-based behavioral intervention program on improving health behavior (dietary intake and physical activity) and anthropometrics of Chinese-American children. A total of 60 children and their families will be recruited. The intervention will include a weekly Internet session tailored to each individual child for eight weeks and three Internet sessions for parents. Children and their parents in the control group will receive general health information on healthy eating, active lifestyles, dental care, smoking cessation, and risk taking issues via the Internet. The content of the sessions is described later. After informed consent is obtained from parents and verbal assent from the children, baseline data (T0) will be collected before assigning the children and parents to the intervention group or control group. Follow-up data for both groups will be collected at 2 months (T1), 4 months (T2) and 6 months (T3) after baseline.

ELIGIBILITY:
Inclusion Criteria:

Children:

* children between the ages of 10 and 14 years old who self-identify as Chinese or of Chinese origin
* reside in the Bay Area in the same household as at least one parent, can read and speak English, and have access to the Internet at home

Parents:

* parents who self-identify as Chinese or of Chinese origin
* have children between the ages of 11 and 14
* are able to read either Chinese or English
* are able to speak Mandarin, Cantonese, or English
* have access to the Internet at home

Exclusion Criteria:

* children with chronic health problems that include any dietary modifications or activity limitations will be excluded (e.g., diabetes, exercise-induced asthma)

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2008-03; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
BMI | baseline to 6 month follow up

SECONDARY OUTCOMES:
physical activity, dietary intake, coping strategy | baseline to 6 month follow up

CONTACTS AND LOCATIONS:
Locations (1):
- University of California San Francisco, San Francisco, California, United States